CLINICAL TRIAL: NCT00317148
Title: Phase II-III Placebo-Controlled, Study to Evaluate the Effects of DHEA on Vasomotor Symptoms (Hot Flashes) in Postmenopausal Women
Brief Title: Effect of Dehydroepiandrosterone (DHEA) on Hot Flashes in Postmenopausal Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-205
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Hot Flashes
Keywords: Hot Flashes; Menopause; Quality of Life; Hot flushes
MeSH Terms: conditions — Hot Flashes | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental)
  Interventions: Drug: Placebos
- DHEA (Experimental)
  Interventions: Drug: DHEA capsule

INTERVENTIONS:
Drug: Placebos — Placebo capsule
  Arms: Placebo
Drug: DHEA capsule — One capsule of DHEA
  Arms: DHEA

SUMMARY:
The purpose of the study is to evaluate the effect of daily oral intake of DHEA 50 mg for 4 months on reducing vasomotor symptoms (hot flashes) compared to placebo administration in postmenopausal women.

DETAILED DESCRIPTION:
Humans, along with the other primates, are unique among animal species in having adrenals that secrete large amounts of the inactive precursor steroids dehydroepiandrosterone (DHEA) and especially its sulfate DHEA-S. The marked reduction in the formation of DHEA-S by the adrenals during aging results in a dramatic fall in the formation of androgens and estrogens in peripheral target tissues, a situation that has been proposed to be associated with age-related diseases including skin atrophy, insulin resistance and obesity. Much attention has been given to the benefits of DHEA administered to postmenopausal women, especially on the bone, skin, vagina and well being after oral as well as percutaneous administration of the precursor steroid.

This study proposes to study the effect of 50 mg oral DHEA capsules during a period of 4 months administered to postmenopausal women experiencing 50 or more moderate to severe hot flushes per week. Participants will be stratified by the number of hot flushes experienced per week. The two strata are: 50-70 or more than 70 hot flushes per week. During the study several biological and clinical parameters will be evaluated, as well as the reduction of the number of hot flashes and improvement of overall quality of life.

Subjects will be evaluated at specific time intervals during the study for the above mentioned parameters as well as tolerability and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women with 50 or more moderate to severe hot flushes.
* Women between 40 to 70 years of age.

Exclusion Criteria:

* Body mass index (BMI) of 35 kg/m2 or more.
* Significant metabolic and endocrine diseases.
* Diagnosis of cancer.
* Use of steroids or drugs that interfere with the metabolism of estrogen.
* Use of any systemic estrogen, progestin, or DHEA in the eight weeks prior to randomization.
* Use of alternative therapies or natural products to treat postmenopausal symptoms in the four weeks prior to randomization.
* Palpable fibroids or uterine prolapse: Grade 2 or 3.
* Cigarette smoking

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2006-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Use of a diary to monitor the number and intensity of hot flashes as compared to placebo at screening, day 1, weeks 2, 4, 8, 12 and 16

SECONDARY OUTCOMES:
Evaluation of safety as well as quality of life, psychological general well being, and sexual life by questionnaires at day 1, 2, 4, 8, 12 and 16 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Leonello Cusan, MD, PhD, Principal Investigator — CHUL Research Center; Fernand Labrie, MD, PhD, Study Director — CHUL Research Director
Locations (1):
- Clinique des Traitements Hormonaux, Sainte-Foy, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arlt W, Callies F, Koehler I, van Vlijmen JC, Fassnacht M, Strasburger CJ, Seibel MJ, Huebler D, Ernst M, Oettel M, Reincke M, Schulte HM, Allolio B. Dehydroepiandrosterone supplementation in healthy men with an age-related decline of dehydroepiandrosterone secretion. J Clin Endocrinol Metab. 2001 Oct;86(10):4686-92. doi: 10.1210/jcem.86.10.7974. PMID 11600526
- [Background] Baulieu EE. Neuroactive neurosteroids: dehydroepiandrosterone (DHEA) and DHEA sulphate. Acta Paediatr Suppl. 1999 Dec;88(433):78-80. doi: 10.1111/j.1651-2227.1999.tb14408.x. PMID 10626550
- [Background] Belanger A, Candas B, Dupont A, Cusan L, Diamond P, Gomez JL, Labrie F. Changes in serum concentrations of conjugated and unconjugated steroids in 40- to 80-year-old men. J Clin Endocrinol Metab. 1994 Oct;79(4):1086-90. doi: 10.1210/jcem.79.4.7962278.
- [Background] Diamond P, Cusan L, Gomez JL, Belanger A, Labrie F. Metabolic effects of 12-month percutaneous dehydroepiandrosterone replacement therapy in postmenopausal women. J Endocrinol. 1996 Sep;150 Suppl:S43-50. PMID 8943786
- [Background] Flynn MA, Weaver-Osterholtz D, Sharpe-Timms KL, Allen S, Krause G. Dehydroepiandrosterone replacement in aging humans. J Clin Endocrinol Metab. 1999 May;84(5):1527-33. doi: 10.1210/jcem.84.5.5672. PMID 10323374
- [Background] Jedrzejuk D, Medras M, Milewicz A, Demissie M. Dehydroepiandrosterone replacement in healthy men with age-related decline of DHEA-S: effects on fat distribution, insulin sensitivity and lipid metabolism. Aging Male. 2003 Sep;6(3):151-6. PMID 14628495
- [Background] Labrie F. Intracrinology. Mol Cell Endocrinol. 1991 Jul;78(3):C113-8. doi: 10.1016/0303-7207(91)90116-a. PMID 1838082
- [Background] Labrie F, Belanger A, Cusan L, Gomez JL, Candas B. Marked decline in serum concentrations of adrenal C19 sex steroid precursors and conjugated androgen metabolites during aging. J Clin Endocrinol Metab. 1997 Aug;82(8):2396-402. doi: 10.1210/jcem.82.8.4160. PMID 9253307
- [Background] Labrie F, Diamond P, Cusan L, Gomez JL, Belanger A, Candas B. Effect of 12-month dehydroepiandrosterone replacement therapy on bone, vagina, and endometrium in postmenopausal women. J Clin Endocrinol Metab. 1997 Oct;82(10):3498-505. doi: 10.1210/jcem.82.10.4306. PMID 9329392
- [Background] Labrie F, Simard J, Luu-The V, Belanger A, Pelletier G, Morel Y, Mebarki F, Sanchez R, Durocher F, Turgeon C, Labrie Y, Rheaume E, Labrie C, Lachance Y. The 3B-hydroxysteroid dehydrogenase/isomerase gene family: lessons from type II 3B-HSD congenital deficiency.In: Signal Transduction in Testicular Cells. Ernst Schering Research Foundation Workshop. Hansson, V., Levy, F.O. and Tasken, K. (eds.), Berlin, Heidelberg, New York, Springer-Verlag, Vol. Suppl. 2:pp. 185-218, 1996.